CLINICAL TRIAL: NCT00346671
Title: Effects of Reiki on Physiological Consequences of Acute Stress
Brief Title: Effects of Reiki on Stress
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Joan Fox, Staff, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R21AT001884-01 (NIH)
Record Dates: First submitted 2006-06-29; First posted 2006-06-30 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Stress
Keywords: Reiki; Stress; CAM
MeSH Terms: interventions — RE1-silencing transcription factor; salicylhydroxamic acid; Touch; Therapeutic Touch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Supine Rest (Placebo Comparator): 30min supine rest listening to soft music
  Interventions: Other: Rest
- Sham Reiki (Sham Comparator): 30 min intervention by sham practitioner
  Interventions: Other: Sham
- Reiki (Experimental): 30 min session with Reiki practitioner
  Interventions: Other: Reiki

INTERVENTIONS:
Other: Rest — 30 min supine rest
  Arms: Supine Rest
Other: Sham — 30 min session with Sham practitioner
  Other Names: Touch; Pretend Reiki; Placebo Reiki
  Arms: Sham Reiki
Other: Reiki — 30 min session with Reiki practitioner
  Other Names: Energy Healing; Energy Therapy; Touch Therapy
  Arms: Reiki

SUMMARY:
Complementary therapies such as Reiki are becoming popular. Reiki is a practice used for relaxation and pain management that involves physical touch and social contact with a trained, empathetic practitioner. Unlike many relaxation therapies, Reiki requires no participation by the patient, a feature that makes Reiki particularly attractive in the hospital setting, where patients are often extremely anxious, depressed, in pain, or sedated. Our primary research questions are to determine whether physiological changes are induced during a Reiki session and whether a Reiki session affects responses to a subsequent acute stressor. Secondary research questions include assessing which benefits result from placebo or unique abilities of "attuned" Reiki practitioners and assessing background characteristics of recipients that are associated with acceptance and responsiveness. Based on its use to reduce pain and anxiety, we will study potential mechanisms by which Reiki decreases activity of the sympathetic nervous system and other stress pathways. Comparison of the responses in a Reiki group with those in supine-control and sham groups will allow us to gain insights into mechanisms by which Reiki effects are mediated. Information obtained from the proposed studies will provide detailed information on physiological pathways affected by Reiki. Should Reiki decrease stress pathways or reduce physiological responses to stressful situations, it could be a useful adjunct to traditional medicine and have significant health and economic benefits.

DETAILED DESCRIPTION:
See Brief Summary

ELIGIBILITY:
Inclusion Criteria:

* Healthy Individuals between the age of 18 and 75

Exclusion Criteria:

* Already involved in regular (one time a week or more) mind-body practices (yoga, meditation, Qi-gong, guided imagery, Taichi, biofeedback; attendance at religious services is not considered a mind-body practice) in the past three months OR has been doing intense spiritual practice for more than 6 months in the past (an average of 6hrs a week)
* Already received an energy therapy treatment (Reiki, therapeutic touch, healing touch, touch therapy) in the past. (note: acupuncture, massage Qi-gong are not considered energy therapies in the context of this study)
* Score on the DASS21 for Depression greater or equal to 21
* Score on the DASS21 for Anxiety greater or equal to 15
* In the last 3 months, has had a major stressful life-event that is likely to affect the outcomes of the study
* Medical condition, current illness or history of chronic illness that might affect the outcomes of the study such as those affecting stress response, cardiovascular, endocrine, or immune systems (Examples: cancer, lupus, multiple sclerosis, blood-clotting disorder, severe allergies or asthma that impairs breathing, diabetes mellitus, hyperglycemia, or hypoglycemia, cardiovascular disease, depression/anxiety etc.)
* In the past 3 months, has used or is chronically using over-the-counter, recreational or prescription drugs that might affect the outcomes of the study such as those affecting cardiovascular, platelets, central nervous system, endocrine, immune systems(Examples: steroid, blood pressure medication, depression/anxiety medication, antiplatelet drugs, etc.)
* Color Blind
* Consume 3 or more alcoholic drinks per day most days over the 3 months
* Pregnant
* Problems donating blood: Fear of hypodermic needles; has felt dizzy or was about to faint following a needle stick
* Incompatibility of energy healing with religious beliefs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2006-01; Primary Completion 2009-10 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
1: To determine whether a Reiki session affects emotional states, ANS, or HPA activity | 3 years
2. To determine whether a Reiki session affects responses to a subsequent acute stressor | 3 years

SECONDARY OUTCOMES:
Assess which benefits result from placebo and which from unique abilities of Reiki practitioners | 3 years
Obtain preliminary information on mechanisms needed for the rational design of a larger clinical trial | 3 years
Assess the role of a variety of baseline variables on responses. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Joan E. Fox, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States